CLINICAL TRIAL: NCT06824324
Title: Is Botulinum Toxin Predictable in the Management of Myofascial Pain Syndrome Related to Masticatory Muscles?
Brief Title: The Use of Botulinum Toxin in the Management of Myofascial Pain Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yassir R. Al-khannaq (Other)
Responsible Party: Sponsor-Investigator, Yassir R. Al-khannaq, LECTURER Dr., University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1004125
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Myofacial Pain Syndrome
MeSH Terms: conditions — Facial Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- injection of Botulinum toxin A in Triger zone (Active Comparator): The method utilized for dilution of Botulinum toxin A involved addition of 2.5ml of normal saline to 100 unit of Botox vial, and addition of 1.25ml to 50U of Botox so each 0.1ml contain 4U of Botox.
  Botox can be denatured easily so the dilution process was very precise and the dilute injected gently in to Botox Vial.
  A thirty units of Botulinum toxin A was injected intramuscularly bilaterally (30 U for each side) in thirteen patients and unilaterally in one patient
  Interventions: Drug: intramuscular Botulinum Toxin

INTERVENTIONS:
Drug: intramuscular Botulinum Toxin — A thirty units of Botulinum toxin A was injected intramuscularly in Triger zone of patient with myofascial pain syndrome

SUMMARY:
The objective of this study was to assess the efficacy of Botulinum toxin type (A) (BoNTA) injection in Myofascial pain syndrome management in the terms of duration of function improvement and pain reduction.

Material and methods: Fourteen patients with Myofascial pain syndrome related to masticatory muscles were presented with trismus, pain and impairment of oral function. Treatment plan was established by utilizing thirty units of Botulinum toxin type (A) which was injected into masseter and sometimes temporalis muscle.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is acute or chronic musculoskeletal pain that characterized by the presence of unique trigger points of pain (TrPs) . Etiology of this condition may include psychogenic stress, prolong muscle strain, trauma to the joint or muscle, arthritis, myositis, chronic infection, and general fatigue. Current therapeutic approaches available for Myofascial pain syndrome involved pharmacological and non-pharmacological treatment options. The non-pharmacological techniques may include a) manual therapy by muscle stretch or massage, b) muscular taut band injection by local anesthesia or botulinum toxin, c) acupuncture, and d) therapeutic ultrasound .

Botulinum toxin is a neurotoxin protein produced by anaerobic bacteria (clostridium botulinum) . It was first discovered by a German physician named Justinus Kerner who observed that the toxin acts by impeding signal transmission in the somatic and autonomic motor systems, leaving the sensory signal transmission uninterrupted .

It blocked the acetylcholine release from the nerve endings thus prevent the neurological signals transmission at the neuromuscular junction. In turn, this reduces the muscle contraction and produces relaxation of the muscle . However, the clinical effects of Botulinum toxin are transit as these neurotoxins degenerate at nerve terminals and became inefficient after a period of time .

Although numerous articles were published on the Botulinum Toxin A (BoNTA) injection in the management of MPS, but there were diverse clinical results in the literature regarding this subject and its effectiveness is still questionable . The objective of this study was to evaluate the efficiency and outcomes of BoNTA injection in the management of MPS related to masticatory muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with myofascial pain related to the muscles of mastication (masseter and temporalis muscle).
2. Patient with regional pain.
3. Patient with or without limited mouth opening (trismus).
4. Presence of trigger points within the identified masticatory muscles.

Exclusion Criteria:

- 1. Hypersensitivity to Botulinum toxin. 2. Active infection in the virtual points of injection. 3. Patient with generalized musculoskeletal pain as in Fibromyalgia Syndrome (FMS).

4. Children younger than 12 years old and pregnant woman. 5-Patient recently undergone to one other modality of treatment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Pain level | 16 weeks
  Pain level was assessed before the initiation of treatment and at 2, 8 and 16 weeks after injection by using the visual analogue scale

SECONDARY OUTCOMES:
Mouth opening | 16 weeks
  Mouth opening was also measured prior and after BoNTA injection by digital caliper. Follow up period was 4 months after the initial injection. Descriptive statics for (pre -post) operative pain and mouth opening at 2 weeks, 16 weeks after injection

CONTACTS AND LOCATIONS:
Locations (1):
- College Of Dentistry University Of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided